CLINICAL TRIAL: NCT04204265
Title: A Prospective Study of a Single Injection Cross-linked Sodium Hyaluronate (MONOVISC) to Provide Symptomatic Relief of Osteoarthritis of Shoulder Joint
Brief Title: MONOVISC for Shoulder Joint Pain Relief Due to Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anika Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MON 18-02
Record Dates: First submitted 2019-12-17; First posted 2019-12-18 (Actual); Results first posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Osteo Arthritis Shoulders
Keywords: Sodium Hyaluronate; Hyaluronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Monovisc (Other): Single injection of Monovisc into the Index Shoulder
  Interventions: Device: Monovisc

INTERVENTIONS:
Device: Monovisc — A chemically cross-linked sodium hyaluronate supplied as a 4 mL unit dose in a 5 mL glass syringe.

SUMMARY:
Obtain real world, post market data to confirm the clinical improvement and safety in patients treated with a single injection of MONOVISC for the symptomatic relief of osteoarthritis in the shoulder joint.

DETAILED DESCRIPTION:
The goal of this study is to demonstrate the clinical improvement and safety in patients treated with MONOVISC for shoulder osteoarthritis. Specifically, this study will provide confirmation to the effectiveness and safety of MONOVISC at relieving shoulder joint pain to 6 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Body Mass Index (BMI) ≤ 45 kg/m2
3. Diagnosis of symptomatic osteoarthritic joint in the index joint (Kellgren Lawrence grade I to III or Guyette grade I to III) to be treated with MONOVISC injection.
4. Failed conservative treatment for joint osteoarthritis.
5. NRS pain ≥4 and ≤9 in the index joint.
6. Subject must be willing to abstain from other treatments of the index joint for the duration of the study.
7. Subject is willing to discontinue all analgesics including NSAIDs, except acetaminophen/paracetamol, at least seven days before the treatment injection and through the completion of the study.
8. Subject is willing to use only acetaminophen/paracetamol (up to a maximum of 4.0 grams per day per the package insert) for the treatment of joint pain for the duration of the study. At least forty-eight hours prior to the Baseline Visit and each follow-up visit, the subject is willing to discontinue use of acetaminophen/paracetamol.
9. Subject is willing to maintain a stable dose of oral glucosamine and/or chondroitin sulfate products throughout the study, if taken prior to signing the informed consent form (ICF).
10. Able and willing to provide signed informed consent.

Exclusion Criteria:

1. History of hypersensitivity to any of the ingredients in the hyaluronan
2. Infection or skin disease in the area of the injection site or index joint
3. NRS pain > 3 in the contralateral joint
4. Subject received an injection of Hyaluronic Acid (HA) and/or steroid in either joint within 6 months of signing the informed consent form (ICF). A subject will be excluded if they are planning to receive an HA or steroid injection (other than the study injection) in either joint during the course of this study.
5. Known inflammatory or autoimmune disorders (including rheumatoid arthritis, gout), or other pre-existing medical conditions that, in the opinion of the investigator, could impact treatment of the index joint or affect the ability of the subject to accurately complete the study questionnaires and comply with the study requirements.
6. Subject is taking medications at the time of signing the ICF which could interfere with the treatment procedure, healing and/or assessments. This includes but is not limited to oral or injectable anticoagulant treatments, anti-aggregant platelet treatment, chronic opioid analgesics. Low dose aspirin used for cardiovascular protection is allowed if a stable regimen is maintained for the duration of the study.
7. Subjects who had an oral, intramuscular, intravenous, rectal suppository or topical (excluded in index joint only) corticosteroid prior 30 days of signing the ICF are excluded. Topical corticosteroid use at any site other than the index joint is allowed.
8. Significant trauma to the index shoulder within 26 weeks of screening
9. Chronic use of narcotics or cannabis.
10. Ligament instability or tear in index joint.
11. Diagnosis of fibromyalgia
12. Diagnosis of osteonecrosis in index joint
13. Uncontrolled diabetes with HbA1c of >7%.
14. Subject is a woman who is pregnant or breastfeeding at the Screening Visit or a woman of child bearing potential who refuses to use effective contraception during the course of the study.
15. Subject is receiving or in litigation for worker's compensation.
16. Otherwise determined by the investigator to be medically unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kara Mezger, Study Director — Anika Therapeutics
Locations (4):
- Krajská zdravotní, a.s., Ústí nad Labem, Czechia
- Poland (3):
  - Nzoz Medi-Spatz, Gliwice
  - SPORTO, Lodz
  - Przychodnia Rodzinna na Sadowej, Torun

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only one shoulder [Index Shoulder] of each participant was included in this study.
Period: Overall Study
Arm/Group | Monovisc
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Monovisc
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.48 (9.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0
Index Shoulder [Count of Participants; unit: Participants]
  Right | 19
  Left | 6

OUTCOME MEASURES:

1. Primary Outcome: Numerical Rating Scale (NRS) Pain
Description: Mean change in Numerical Rating Scale (NRS) Pain in the Index Shoulder from baseline to 6 Months post injection. NRS is an 11-Point scale where 0=No Pain, 10=Worst Pain. A larger negative value (maximum -10.0) for the change from baseline indicates less pain and a better clinical outcome following treatment.
Time Frame: From Baseline to 6 Months
Population: Intent To Treat (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Monovisc
Number analyzed (Participants) | 25
score on a scale | -4.12 (2.21)
Statistical Analysis 1: Comparison: Monovisc; Test type: Other; p < 0.0001, t-test, 1 sided — P-Value was calculated

2. Secondary Outcome: Disabilities of Arm, Shoulder & Hand (DASH) Index
Description: Mean change in the Index Shoulder Disabilities of the Arm, Shoulder and Hand (DASH) Index from baseline to 6 months post injection. The DASH Index is a 30-item self-reported questionnaire on pain and function in which the response options are presented as 5-point Likert scales. Scores for each question range from 0=(no pain or disability) to 100=(most severe pain or disability) and are averaged to calculate the final DASH Index score.
  A negative value for the change in DASH Index score indicates improvement.
  A larger negative value indicates a higher level of improvement, and a better clinical outcome.
Time Frame: From Baseline to 6 Months
Population: Intent To Treat (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Monovisc
Number analyzed (Participants) | 25
score on a scale | -36.22 (17.43)
Statistical Analysis 1: Comparison: Monovisc; Test type: Other; p < 0.0001, t-test, 1 sided — P-Value was calculated

3. Secondary Outcome: Patient Global Assessment (PGA) Score
Description: Mean change from baseline to 6 months in Index Shoulder pain post treatment as measured by the Patient Global Assessment (PGA) Score. PGA Score records participant responses to their assessment of how much their STUDY (treated) shoulder is bothering them today . The PGA Score is a validated 11-point Likert scale from 0=No Pain to 10=Worst Pain.
  A negative value for the change from baseline indicates improvement in PGA Score. A larger negative value (maximum -10.0) for the change from baseline indicates less pain and a better clinical outcome following treatment.
Time Frame: From Baseline to 6 Months
Population: Intent To Treat (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Monovisc
Number analyzed (Participants) | 25
score on a scale | -4.16 (2.36)
Statistical Analysis 1: Comparison: Monovisc; Test type: Other; p < 0.0001, t-test, 1 sided — P-Value was calculated

4. Secondary Outcome: The Outcomes Measures for Rheumatic Arthritis Clinical Trials-Osteoarthritis Research Society International (OMERACT-OARSI) Responder Index
Description: The post-treatment responder rate at 6 months as determined through a calculation defined by the Outcomes Measures for Rheumatic Arthritis Clinical Trials-Osteoarthritis Research Society International (OMERACT-OARSI) Responder Index. The OMERACT-OARSI Responder Index reports the percentage of subjects that met the criteria to be a good responder to treatment.
  The criteria for response are (1) improvement in pain or physical function >50% and an absolute change >20 mm; or (2) improvement of >20% with an absolute change >10 mm in at least of the following three categories: pain, physical function, and patient's global assessment.
  A higher percentage of subjects responding to treatment indicates better clinical outcomes.
Time Frame: 6 Months
Population: Intent To Treat (ITT)
Measure: Count of Participants; unit: Participants
Arm/Group | Monovisc
Number analyzed (Participants) | 25
Participants | 23

5. Secondary Outcome: Number of Participants NOT Using Rescue Medication (Acetaminophen/Paracetamol)
Description: The usage of Rescue Medication (RM) at 6 months post treatment as based on the number of participants that were NOT using acetaminophen/paracetamol RM for pain or discomfort.
  A larger percentage of participants that were NOT using RM may correlate to a better clinical outcome in terms of pain.
Time Frame: 6 Months
Population: Intent To Treat (ITT)
Measure: Count of Participants; unit: Participants
Arm/Group | Monovisc
Number analyzed (Participants) | 25
Participants | 21

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the time of the Baseline Study Visit until Study Completion at 26 Weeks (6 months).
Description: The definitions of adverse events and serious adverse events is the same as used in the clinicaltrials.gov definitions.
  The incidence, timing, severity, and relationship to treatment of all Adverse Events (AE) were collected and coded using Medical Dictionary for Regulatory Activities (MedDRA).
Arm/Group | Monovisc
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 5/25
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Monovisc (N=25)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (2)
Hypertension (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
There were no limitations or caveats associated with the conduct of this trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
INVESTIGATOR may publish the Data/Results with the consent of the SPONSOR if:

1. Publication is done after primary publication covering data from all participating sites, and provided the Data/Results do not contain any Confidential Information.
2. Eighteen (18) months has elapsed after entire completion of the Clinical Trial at all participating sites.

DOCUMENTS (2):
  • Study Protocol (2019-08-14): https://cdn.clinicaltrials.gov/large-docs/65/NCT04204265/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-09): https://cdn.clinicaltrials.gov/large-docs/65/NCT04204265/SAP_001.pdf